CLINICAL TRIAL: NCT03749239
Title: Effect of Intake of Enzymatically Hydrolyzed and Non-enzymatically Hydrolyzed Collagen Protein on the Amino Acid Profile of the Blood
Brief Title: Effects of Collagen Protein on the Amino Acid Profile of the Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Collagen_2018
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2018-11

CONDITIONS: Collagen Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effects of collagen protein. (Experimental): Non-hydrolized collagen protein
  Interventions: Dietary Supplement: Collagen protein

INTERVENTIONS:
Dietary Supplement: Collagen protein — Collagen protein

SUMMARY:
This project aims to investigate the absorption of enzymatically hydrolysed and non-enzymatically hydrolysed collagen on the Amino acid profile of the blood

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Medicine influencing protein turnover
* Diabetes
* Smoking

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Amino acid profile of the blood | Blood samples is collected at pre, 0 min, 20 min, 40 min, 60 min, 90 min, 120 min, 180 min and 240 min.
  AA concentrations in blood samples is determined using 1H NMR spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark